CLINICAL TRIAL: NCT00011726
Title: Lead Mobilization & Bone Turnover in Pregnancy/Lactation
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 7437-CP-001
Record Dates: First submitted 2001-02-27; First posted 2001-03-01 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Lead Poisoning
Keywords: Pregnancy; Lead Exposure; Lactation; Bone Mineralization; Maternal-Fetal Exchange
MeSH Terms: conditions — Lead Poisoning; Breast Feeding

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
We are examining the role of maternal bone lead turnover during pregnancy and lactation as a potential source of lead exposure for the fetus and the infant (via breast milk). A cohort, ascertained at entry to care, consists of >1000 women to be followed through pregnancy. In the postpartum subjects are recruited for a nested case control study to assess the influence of lactation on maternal bone density, maternal blood lead and breast milk lead.

ELIGIBILITY:
1. Positive pregnancy test, age 12-35 and informed consent;
2. Gestation <28 weeks at entry to prenatal care;
3. No history of serious chronic or metabolic diseases, which could affect maternal growth or bone density;
4. Not corticosteroid user or diagnosed use of illicit drugs;
5. Eligible for lactation study: Ascertainment during or participation in the pregnancy study and a negative pregnancy test.

Ages: 12 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000
Dates: Start 1996-08; Study Completion 2002-12

REFERENCES:
- [Background] Sowers M, Jannausch M, Scholl T, Schall J. The reproducibility of ultrasound bone measures in a triethnic population of pregnant adolescents and adult women. J Bone Miner Res. 1998 Nov;13(11):1768-74. doi: 10.1359/jbmr.1998.13.11.1768. PMID 9797487
- [Background] Sowers MF, Scholl T, Harris L, Jannausch M. Bone loss in adolescent and adult pregnant women. Obstet Gynecol. 2000 Aug;96(2):189-93. doi: 10.1016/s0029-7844(00)00903-0. PMID 10908761
- [Background] Scholl TO. High third-trimester ferritin concentration: associations with very preterm delivery, infection, and maternal nutritional status. Obstet Gynecol. 1998 Aug;92(2):161-6. doi: 10.1016/s0029-7844(98)00157-4. PMID 9699743
- [Background] Goodlin RC. High third-trimester ferritin concentration: associations with very preterm delivery, infection, and maternal nutritional status. Obstet Gynecol. 1999 Jan;93(1):156. doi: 10.1016/s0029-7844(98)00427-x. No abstract available. PMID 9916975
- [Background] Scholl TO. Teenage pregnancy. In "Cambridge Encyclopedia of Growth and Development", SJ Ulijaszek, FE Johnson, MA Preece (eds), Cambridge Univ Press, 312-13,1998
- [Background] Scholl TO, Reilly T. Essential trace elements and mineral nutrition in human pregnancy. In "Clinical nutrition of the essential trace elements and mineral - The Guide for Health Professionals", John R. Bogden, Leslie Klevay (eds), Humana Press, 1999. ( In press)